CLINICAL TRIAL: NCT05020028
Title: The Use of Cannabidiol (CBD) in Pain Reduction for Knee Osteoarthritis. A Double-Blind, Randomized Control Study
Brief Title: Cannabidiol (CBD) in Pain Reduction for Knee Osteoarthritis
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Orcosa Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 21-00334
Record Dates: First submitted 2021-07-13; First posted 2021-08-25 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Knee Arthritis
MeSH Terms: interventions — Cannabidiol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CBD Group (Experimental): The first cohort will take two 25mg cannabidiol (total dose: 50mg) Orally Disintegrating Tablets (CBD ODT) three times daily for a maximum dose of 150mg per day.
  Interventions: Drug: Cannabidiol (CBD)
- Placebo Group (Placebo Comparator): Cohort 2 will receive the same instructions, but with the placebo Orally Disintegrating Tablets (ODT) instead.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cannabidiol (CBD) — Patients will be dispensed enough 25mg cannabidiol (CBD) Orally Disintegrating Tablets (ODT) to take a standard dose of 50mg three times daily for 84 days.
  Other Names: Cannabidiol
  Arms: CBD Group
Drug: Placebo — 25mg Placebo ODT looks like the cannabidiol (CBD) Orally Disintegrating Tablets (ODT), but contains no active ingredients.
  Arms: Placebo Group

SUMMARY:
The purpose of this study is to see if cannabidiol (CBD) orally dissolving tablets (ODTs) can lessen pain, improve function, and improve patient satisfaction in cases of knee osteoarthritis. CBD comes from the cannabis plant and is non-psychoactive (i.e. does not produce a 'high' or altered mental state) as compared to tetrahydrocannabinol (THC), another compound found in cannabis. Researchers are studying different forms of CBD for potential use in treating pain, inflammation, and illnesses.

DETAILED DESCRIPTION:
This will be a multi-center, double-blinded, randomized, placebo-controlled study. The study is comparing pain, outcomes, and patient satisfaction in two cohorts: patients with knee OA undergoing physiotherapy/home exercises who receive CBD and a placebo group with PT/home exercise program. Patients will be asked on treatment Day 1, 2, 7, and 14, 28, 42, and 84 to rate their pain according to the VAS scale. Additionally, patient satisfaction and clinical outcomes will be measured.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting with knee osteoarthritis (KL Grade II-III)
* Knee pain for at least three months, occurring in at least half of the days in that period
* VAS ≥ 4
* Patients ages 40-75, inclusive
* If female patients are pre-menopausal they must be currently practicing effective forms of two types of birth control, which are defined as those, alone or in combination, that result in a low failure rate (less than 1% per year) when used consistently and correctly
* Male patients must be using an effective form of contraception

Exclusion Criteria:

* Knee Injections within the last 3 months (cortisone, PRP, hyaluronic acid)
* Legally incompetent or mentally impaired (e.g., minors, Alzheimer's subjects, dementia, etc.)
* Younger than 40 years of age
* Older than 75 years of age
* Any patient considered a vulnerable subject: pregnant women or fetuses, children, cognitively impaired adults, prisoners
* History of cannabis abuse or dependence
* History of coagulation abnormalities and thromboembolic disease or current abnormal coagulation test values
* History of stroke or acute coronary syndromes within 3 months
* Abnormal coagulation profile
* Renal failure (serum creatinine > 250 μmol/L [2.83 mg/dL]) or liver cirrhosis
* Patients that have been on opioid management for any reason just prior to the study
* Patients with known inflammatory arthritis (such as rheumatoid arthritis, gout, pseudogout etc)
* Patients with a large effusion
* Patients with a BMI > 35
* Patients meeting the DSM-V for major psychiatric illness, such as bipolar disorder
* Patients diagnosed with major depression, psychosis, or substance abuse disorder
* Patients with current or a history of suicidal ideation
* Breastfeeding females
* Abnormal LFTs
* Patients with major neurological disorders, such as dementia, Parkinson's disease, cognitive impairment, epilepsy, history of traumatic brain/head injury, or seizures
* Patients with moderate (Child-Pugh B) and severe hepatic impairment (Child-Pugh C).
* Patients taking moderate or strong inhibitors of CYP3A4 and CYP2C19 (listed below) concomitantly will be considered for exclusion if determined to be clinically significant by the treating physicians
* Patients taking strong CYP3A4 and CYP2C19 inducers (listed below) concomitantly will be considered for exclusion if determined to be clinically significant by the treating physicians
* Patients taking substrates of UTG1A9, UTGB17, CYP2A1, CYP2B6, CYP2C8, CYP2C9 and CYP2C19 (listed below) concomitantly will be considered for exclusion if determined to be clinically significant by the treating physicians

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-06-22 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
VAS Pain Severity Score | Day 1
  A Visual Analogue Scale (VAS) will be used to measure differences in pain between patients receiving CBD with knee OA undergoing physiotherapy compared to patients who do not receive CBD. Patients rate their pain on a scale ranging from 0 (no pain) to 10 (worst pain imaginable). Total scores range from 0-10; higher scores indicates greater pain intensity.
VAS Pain Severity Score | Day 2
  A Visual Analogue Scale (VAS) will be used to measure differences in pain between patients receiving CBD with knee OA undergoing physiotherapy compared to patients who do not receive CBD. Patients rate their pain on a scale ranging from 0 (no pain) to 10 (worst pain imaginable). Total scores range from 0-10; higher scores indicates greater pain intensity.
VAS Pain Severity Score | Day 7
  A Visual Analogue Scale (VAS) will be used to measure differences in pain between patients receiving CBD with knee OA undergoing physiotherapy compared to patients who do not receive CBD. Patients rate their pain on a scale ranging from 0 (no pain) to 10 (worst pain imaginable). Total scores range from 0-10; higher scores indicates greater pain intensity.
VAS Pain Severity Score | Day 14
  A Visual Analogue Scale (VAS) will be used to measure differences in pain between patients receiving CBD with knee OA undergoing physiotherapy compared to patients who do not receive CBD. Patients rate their pain on a scale ranging from 0 (no pain) to 10 (worst pain imaginable). Total scores range from 0-10; higher scores indicates greater pain intensity.
VAS Pain Severity Score | Day 28
  A Visual Analogue Scale (VAS) will be used to measure differences in pain between patients receiving CBD with knee OA undergoing physiotherapy compared to patients who do not receive CBD. Patients rate their pain on a scale ranging from 0 (no pain) to 10 (worst pain imaginable). Total scores range from 0-10; higher scores indicates greater pain intensity.
VAS Pain Severity Score | Day 42
  A Visual Analogue Scale (VAS) will be used to measure differences in pain between patients receiving CBD with knee OA undergoing physiotherapy compared to patients who do not receive CBD. Patients rate their pain on a scale ranging from 0 (no pain) to 10 (worst pain imaginable). Total scores range from 0-10; higher scores indicates greater pain intensity.
VAS Pain Severity Score | Day 84
  A Visual Analogue Scale (VAS) will be used to measure differences in pain between patients receiving CBD with knee OA undergoing physiotherapy compared to patients who do not receive CBD. Patients rate their pain on a scale ranging from 0 (no pain) to 10 (worst pain imaginable). Total scores range from 0-10; higher scores indicates greater pain intensity.

SECONDARY OUTCOMES:
Knee Injury and Osteoarthritis Outcome Score (KOOS) | Baseline
  KOOS is a knee-specific instrument, developed to assess patients' opinion about their knee and associated problems. The five patient-relevant subscales of KOOS are scored separately: Pain (9 items); Symptoms (7 items); ADL Function (17 items); Sport and Recreation Function (5 items); Quality of Life (4 items).
  Patients rank each item using a 5-piont Likert scale ranging from 0 (No Problems) to 4 (Extreme Problems) and each of the five scores are calculated as the sum of the items included. Scores are transformed to a 0-100 scale, with zero representing extreme knee problems and 100 representing no knee problems.
Knee Injury and Osteoarthritis Outcome Score (KOOS) | Week 6
  KOOS is a knee-specific instrument, developed to assess patients' opinion about their knee and associated problems. The five patient-relevant subscales of KOOS are scored separately: Pain (9 items); Symptoms (7 items); ADL Function (17 items); Sport and Recreation Function (5 items); Quality of Life (4 items).
  Patients rank each item using a 5-piont Likert scale ranging from 0 (No Problems) to 4 (Extreme Problems) and each of the five scores are calculated as the sum of the items included. Scores are transformed to a 0-100 scale, with zero representing extreme knee problems and 100 representing no knee problems.
Knee Injury and Osteoarthritis Outcome Score (KOOS) | Week 12
  KOOS is a knee-specific instrument, developed to assess patients' opinion about their knee and associated problems. The five patient-relevant subscales of KOOS are scored separately: Pain (9 items); Symptoms (7 items); ADL Function (17 items); Sport and Recreation Function (5 items); Quality of Life (4 items).
  Patients rank each item using a 5-piont Likert scale ranging from 0 (No Problems) to 4 (Extreme Problems) and each of the five scores are calculated as the sum of the items included. Scores are transformed to a 0-100 scale, with zero representing extreme knee problems and 100 representing no knee problems.
Knee Injury and Osteoarthritis Outcome Score (KOOS) | Week 60
  KOOS is a knee-specific instrument, developed to assess patients' opinion about their knee and associated problems. The five patient-relevant subscales of KOOS are scored separately: Pain (9 items); Symptoms (7 items); ADL Function (17 items); Sport and Recreation Function (5 items); Quality of Life (4 items).
  Patients rank each item using a 5-piont Likert scale ranging from 0 (No Problems) to 4 (Extreme Problems) and each of the five scores are calculated as the sum of the items included. Scores are transformed to a 0-100 scale, with zero representing extreme knee problems and 100 representing no knee problems.
VAS Satisfaction with Pain Management Score | Day 1
  A Visual Analogue Scale (VAS) will be used to measure patient satisfaction with pain management. Patients rate their satisfaction on a scale ranging from 0 (no satisfaction) to 10 (as satisfied as possible). Total scores range from 0-10; higher scores indicates greater satisfaction with pain management.
VAS Satisfaction with Pain Management Score | Day 2
  A Visual Analogue Scale (VAS) will be used to measure patient satisfaction with pain management. Patients rate their satisfaction on a scale ranging from 0 (no satisfaction) to 10 (as satisfied as possible). Total scores range from 0-10; higher scores indicates greater satisfaction with pain management.
VAS Satisfaction with Pain Management Score | Day 7
  A Visual Analogue Scale (VAS) will be used to measure patient satisfaction with pain management. Patients rate their satisfaction on a scale ranging from 0 (no satisfaction) to 10 (as satisfied as possible). Total scores range from 0-10; higher scores indicates greater satisfaction with pain management.
VAS Satisfaction with Pain Management Score | Day 14
  A Visual Analogue Scale (VAS) will be used to measure patient satisfaction with pain management. Patients rate their satisfaction on a scale ranging from 0 (no satisfaction) to 10 (as satisfied as possible). Total scores range from 0-10; higher scores indicates greater satisfaction with pain management.
VAS Satisfaction with Pain Management Score | Day 28
  A Visual Analogue Scale (VAS) will be used to measure patient satisfaction with pain management. Patients rate their satisfaction on a scale ranging from 0 (no satisfaction) to 10 (as satisfied as possible). Total scores range from 0-10; higher scores indicates greater satisfaction with pain management.
VAS Satisfaction with Pain Management Score | Day 42
  A Visual Analogue Scale (VAS) will be used to measure patient satisfaction with pain management. Patients rate their satisfaction on a scale ranging from 0 (no satisfaction) to 10 (as satisfied as possible). Total scores range from 0-10; higher scores indicates greater satisfaction with pain management.
VAS Satisfaction with Pain Management Score | Day 84
  A Visual Analogue Scale (VAS) will be used to measure patient satisfaction with pain management. Patients rate their satisfaction on a scale ranging from 0 (no satisfaction) to 10 (as satisfied as possible). Total scores range from 0-10; higher scores indicates greater satisfaction with pain management.
Number of Patients Requiring Rescue Corticosteroid Use | Up to Week 60

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Alaia, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
The data will only be available to the researchers involved in this study.